CLINICAL TRIAL: NCT04935957
Title: Study of GLUCUBE Performance, a Non-invasive System for Monitoring Blood Glucose Levels Based on Near Infrared Spectroscopy (NIRS) Technology.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: iGluco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DIA-2021-01
Record Dates: First submitted 2021-06-04; First posted 2021-06-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Blood Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non-interventional. Open Label. (Other): GLUCUBE system performance in the monitoring and measurement of the blood glucose compared to the standard glucometer (blood capillary glucometer - Bayer Contour®Next).
  Interventions: Device: GLUCUBE device

INTERVENTIONS:
Device: GLUCUBE device — device to monitor and measure the blood glucose compared to the standard glucometer in a group subjects
  Other Names: GLUCUBE

SUMMARY:
This study is a prospective, single center, non-interventional, open label clinical investigation. The primary objective of the study is to evaluate the performance of GLUCUBE system compared to the standard glucometer in the determination of blood glucose level in adult patients.

DETAILED DESCRIPTION:
The current methods for blood glucose measurements, glucometers, although minimally invasive, can be painful, requiring puncturing the fingertip with a lancet device and removing a drop of blood, that applies to a disposable test strip. This minimal invasiveness may cause discomfort and deter the user from measuring his/her blood glucose levels as frequently as required. Due to GLUCUBE device non-invasive nature, it is expected to give the patient or health care provider immediate reliable quantitative as well as qualitative information, safely and painlessly avoiding any type of discomfort to the user.

This study is a prospective, single center, non-interventional, open label clinical investigation designed with a total amount of 105 subjects. Study participants will take the GLUCUBE device and standard glucometer home and each subject will take 4 pairs of measurements per day for a week.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18 years old.
2. Have a smartphone with an internet connection that allows the installation of GLUCUBE APP
3. Have signed the informed consent.

Exclusion Criteria:

1. Subject is currently participating in another clinical investigation or has participated in another clinical investigation in the past 30 days prior to the start of the present study.
2. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period.
3. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
4. Patients with any acute active and/or infectious disease.
5. Patients who have a condition that affects blood circulation in the fingers of the hand, such as Raynaud's phenomenon.
6. Any medical condition that, by the investigator judgment, will increase the risk from hyper and hypoglycemic event: seizures, heart disease, hypoglycemia unawareness, etc.
7. Patients who, in the opinion of the investigator, do not have sufficient manual dexterity to perform the tests themselves.
8. Patients with an inability to maintain stability of the hand during measurement or with progressive disease of the nervous system that affects movement (Parkinson's disease, moderate-severe essential tremor, and other diseases with involuntary movements).
9. Patients suffering from calluses, malformations, or open wounds with bandages.
10. Patients with nail polish or any type of false nail.
11. Subjects who do not understand or cannot follow the Procedures Involved in the Use of the Device Under Investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Performance Evaluation | 4 times/day for 1 week
  GLUCUBE system performance in the monitoring and measurement of the blood glucose compared to the standard glucometer (blood capillary glucometer - Bayer Contour®Next).
  Each pair of measurements includes one measurement with the standard glucometer (Bayer Contour®Next) and one measurement with GLUCUBE device.
Safety Evaluation | All AE will be collected during participation in the study since V1 at V2 (8 days)
  All (Serious) Adverse Events and GLUCUBE device related adverse events: local and systemic effects of GLUCUBE device, and the standard glucometer, including, but not limited to redness, burns, pain, or other complications such as bleeding or local infection will be collected.

SECONDARY OUTCOMES:
Performance Evaluation | through study completion, an average of 8 days
  GLUCUBE system performance in the monitoring and measurement of the blood glucose compared to the standardized POC device for the determination of glucose (Accu-Chek® Inform II system).
  Each pair of measurements includes one measurement with standardized POC device for the determination of glucose (Accu-Chek® Inform II system) and one measurement with GLUCUBE device.

OTHER OUTCOMES:
User satisfaction | 8 days after the participant enters the study
  Patient reported satisfaction related to the investigational device: in a 1 to 10 scale: 1 - Disagree, 10 - Agree.
  And, if given the choice, will you use GLUCUBE device again? Yes or No

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Salud La Algaba, La Algaba, Sevilla, Spain